CLINICAL TRIAL: NCT05650086
Title: A Phase II Study to Evaluate Accuracy of ThermalytixTM in Detecting Breast Cancer
Brief Title: Novel Thermal Imaging Technique for Breast Screening
Status: Terminated | Type: Observational
Why Stopped: PI has left the institution (University of Arizona Cancer Center).
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00001233
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Thermal Imaging; Artificial Intelligence; Breast Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Biopsy: Subjects who are scheduled for biopsy will be enrolled.
  Interventions: Device: Thermalytix
- Cohort 2: Screening mammogram: Patients who underwent screening mammogram will be enrolled.
  Interventions: Device: Thermalytix
- Cohort 3: Diganostic mammogram: Subjects scheduled for diagnostic mammogram will be enrolled.
  Interventions: Device: Thermalytix
- Cohort 4: Prior history of lympectomy, routine mammogram: Subjects with prior history of lumpectomy scheduled for their routine mammogram will be enrolled.
  Interventions: Device: Thermalytix

INTERVENTIONS:
Device: Thermalytix — One-time Thermal imaging is performed for this cohort.

SUMMARY:
This trial is to study a new breast imaging tool called Thermalytix™. ThermalytixTM is a new radiation-free, automated breast cancer screening technique that uses Artificial Intelligence (AI) over thermal images. Thermal images are heat signatures in our body. This new technique will capture heat signatures in the breast and analyze those images with AI software. This study will evaluate the performance of ThermalytixTM breast imaging against standard imaging modalities, such as mammography and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Be capable of understanding the investigational nature of the study and all pertinent aspects of the study
* Be capable of signing and providing written consent in accordance with institutional and federal guidelines
* Be willing and able to comply with scheduled visits, treatment plan, and follow up with research staff
* Age ≥ 21 years
* Cohort specific criteria
* Cohort 1: Be scheduled for biopsy
* Cohort 2: Had a normal screening mammogram within 3 months of study enrollment
* Cohort 3: Be scheduled for diagnostic mammogram
* Cohort 4: History of breast cancer, s/p lumpectomy and be scheduled for routine mammogram

Exclusion Criteria:

* Cohort specific criteria
* Cohort 1: Previous biopsies in the same or opposite breast within 3 months of study enrollment, prior history of breast cancer, prior history of breast surgeries including implants
* Cohort 2: prior history of breast surgeries including implants
* Cohort 3: Already underwent a biopsy in the same or opposite breast within 3 months of study enrollment, prior history of breast cancer, prior history of breast surgeries including implants
* Cohort 4: surgery <1 year, h/o mastectomy with reconstruction
* Unable to complete study related procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for breast biopsy or mammogram
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of ThermalytixTM in detecting breast cancer | Through study completion, an average of 30 days
  Determine sensitivity and specificity of ThermalytixTM in detecting breast cancer in patients scheduled to undergo breast biopsy (Cohort 1). The sensitivity and specificity will be estimated using 95% exact binomial confidence intervals. The required sample size was determined based on the target sensitivity and specificity, and the resulting confidence intervals.

SECONDARY OUTCOMES:
Sensitivity and specificity of ThermalytixTM in assessing need for biopsy | Through study completion, an average of 30 days
  To determine accuracy of ThermalytixTM in assessing need for biopsy in patients who are found to have abnormal screening mammogram. Cohort 1 subjects will be used to determine this endpoint. The sensitivity and specificity will be estimated using 95% exact binomial confidence intervals. The required sample size was determined based on the target sensitivity and specificity, and the resulting confidence intervals.
Correlate normal screening mammogram results with ThermalytixTM results | Through study completion, an average of 30 days
  To compare ThermalytixTM with screening mammogram in healthy subjects undergoing routine screening. Cohort 2 will be used to assess this endpoint. The specificity will be estimated using 95% exact binomial confidence intervals. The required sample size was determined based on the target specificity, and the resulting confidence intervals.
Correlate diagnostic mammogram results with ThermalytixTM results | Through study completion, an average of 30 days
  To compare ThermalytixTM with diagnostic mammogram in subjects who underwent diagnostic mammogram. Cohort 3 will be used for this endpoint. The specificity will be estimated using 95% exact binomial confidence intervals. The required sample size was determined based on the target specificity, and the resulting confidence intervals.
Correlate mammogram results with ThermalytixTM results in patients who underwent lumpectomy | Through study completion, an average of 30 days
  To compare ThermalytixTM with mammogram result (screening or diagnostic) in women who underwent lumpectomy. Cohort 4 will be used for this endpoint. The specificity will be estimated using 95% exact binomial confidence intervals. The required sample size was determined based on the target specificity, and the resulting confidence intervals.
Report patient experience with ThermalytixTM | Through study completion, an average of 30 days
  Patient experience with ThermalytixTM will be documented via questionnaires. On a scale of 1-5, patients will document their experience during their mammogram and Thermalytix exam; in general, higher values indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No